CLINICAL TRIAL: NCT01658371
Title: Preference of CYP450 2B6 516 G>T Polymorphism and Pharmacokinetics of Plasma Efavirenz in A Group of HIV Infected Southern Chinese
Brief Title: Preference of Genetic Polymorphism and Pharmacokinetics
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, To Kin Wang, Specialist, Chinese University of Hong Kong
Other Study IDs: CRE-2008.180
Record Dates: First submitted 2012-02-27; First posted 2012-08-07 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: HIV
Keywords: HIV

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- efavirenz: HIV patients on efavirenz

SUMMARY:
Genetic polymorphism affects plasma concentration of antiretroviral therapy in HIV patients. The investigators investigate the prevalence of genetic polymorphism affecting efavirenz metabolism and the corresponding pharmacokinetics of different genotypes.

DETAILED DESCRIPTION:
Eligible patients are invited to donate blood samples for pharmacokinetic study and genotype analysis

ELIGIBILITY:
Inclusion Criteria:

* Southern Chinese HIV patients on efavirenz

Exclusion Criteria:

* Refuse to sign consent, HIV patients not on efavirenz

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Southern Chinese HIV patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics | 24 hour
  This includes plasma concentration of drugs in relation to time, in different genotypes

SECONDARY OUTCOMES:
genotypes frequency | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: S S Lee, Professor, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong, China